CLINICAL TRIAL: NCT03723343
Title: Prospective Phase II Clinical Study of GP-induced Chemotherapy Combined With IMRT and TPF-induced Chemotherapy Combined With IMRT in the Treatment of Nasopharyngeal Carcinoma
Brief Title: GP-induced Chemotherapy Combined With IMRT and TPF-induced Chemotherapy Combined With IMRT in the Treatment of Distant Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Feng Jing, Head and neck cancer director, chief researcher, clinical professor, Guiyang Medical University
Other Study IDs: 201805045
Record Dates: First submitted 2018-10-18; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Experimental: GP+IMRT: Test group: GP-induced chemotherapy (Gemcitabine 1000 mg/m2 d1, 8+Cisplatin 80 mg/m2 d1, once every 3 weeks, 4/6 course) + IMRT radiotherapy alone
  Interventions: Drug: GP+IMRT
- Active Comparator: TPF+IMRT: Control group: TPF-induced chemotherapy (Docetaxel: 75 mg/m2d1, Cisplatin 75 mg/m2, d1~d5, 5-fluorouracil 750 mg/m2/dd1~d5, 4/6 course) + IMRT radiotherapy alone
  Interventions: Drug: TPF+IMRT

INTERVENTIONS:
Drug: GP+IMRT — Gemcitabine 1000 mg/m2 intravenously, d1&d8 +Cisplatin 80 mg/m2 intravenously, d1 21~28 days/cycle, 4 patients with oligometastasis, 6 cycles with multiple metastases
  Other Names: Experimental group
  Groups: Experimental: GP+IMRT
Drug: TPF+IMRT — Docetaxel: 75mg/m2 intravenous drip, d1+Cisplatin75mg/m2 intravenous drip, d1~d5+5-fluorouracil 750mg/m2/d intravenous drip, d1~d521~28 days/cycle, patients with oligometastasis take 4 cycles, moreTransfer patients for 6 cycles
  Other Names: Control group
  Groups: Active Comparator: TPF+IMRT

SUMMARY:
Mainly compared with GP induction chemotherapy combined with IMRT and TPF induction chemotherapy combined with IMRT in the treatment of nasopharyngeal carcinoma, the cure rate, remission rate, treatment of distant metastases and lymph node metastasis, quality of life improvement rate, etc.

DETAILED DESCRIPTION:
1. The main purpose: Whether the GP program can improve the efficiency of patients with nasopharyngeal carcinoma, especially overall survival (OS), in the TPF program. 2. Secondary purpose: To compare the progression-free survival (PFS) local failure-free survival (LR-FFS), the short-term remission rate of the tumor, the adverse chemotherapy response, and the treatment compliance Sex, as well as quality of life. 3. Significance of the research project Nasopharyngeal carcinoma is sensitive to radiotherapy and chemotherapy. Platinum-based chemotherapy is used in the treatment of distant metastasis and metastasis. It can effectively alleviate local symptoms and reduce local symptoms. The tumor volume thereby reduces the high dose area of the target area. Primary lesions and lymphatic drainage area radiotherapy can reduce tumor burden, relieve symptoms, and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. The pathological type is non-keratinized cancer (according to the pathological classification of the World Health Organization, WHO).
2. The stage is TxNxM1 (according to the eighth edition of the AJCC staging standard) (Appendix I).
3. There is evidence of distant transfer (M1).
4. functional status: Karnofsky scale (KPS) > 70 (Appendix II).
5. normal bone marrow function: white blood cell count > 4 × 109 / L, hemoglobin > 90g / L and platelet count > 100 × 109 / L.
6. normal liver function: alanine aminotransferase (ALT), aspartate aminotransferase (AST) <1.5 times the upper limit of normal (ULN), and alkaline phosphatase (alkaline phosphatase, ALP) < 2.5 x ULN and bilirubin < ULN.
7. normal renal function: creatinine clearance (creatinine clearance) > 60 ml / min.
8. The patient must be informed of the basic content of the study and sign an informed consent form.

   -

Exclusion Criteria:

1. the pathological type is WHO keratinized squamous cell carcinoma or basal squamous cell carcinoma.
2. age > 65 years old or < 18 years old.
3. a history of malignant tumors, except for adequately treated basal cell carcinoma or squamous cell carcinoma and cervical carcinoma in situ.
4. Women during pregnancy or lactation (pregnancy tests should be considered for women of childbearing age; effective contraception should be emphasized during treatment).
5. has received radiation therapy (if it is non-melanoma skin cancer and the previous lesion is placed

   Except for the target area of treatment.
6. primary lesions and cervical metastases have received chemotherapy or surgery (except for diagnostic treatment).
7. accompanied by other serious diseases, may bring greater risk or affect the compliance of the test. For example: unstable heart disease, kidney disease, chronic hepatitis, uncontrolled diabetes (fasting blood glucose > 1.5 x ULN), and mental illness. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nasopharyngeal carcinoma with a distance between 18 and 65
Sampling Method: Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2018-10-18 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 3 years
  Progress-free survival(year) is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  The OS(year) was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional failure-free survival(LRFS) | 3 years
  The LRFS(year) is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant metastasis-free survival(DMFS) | 3 years
  The DMFS(year) is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Overall response rate | 3 years
  Tumour response(CR/PR/SD/PD) was classified according to RECIST v1.1
Incidence of acute and late toxicity | 3 years
  Incidence of acute toxicity（Grade1/2/3/4） is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Long, Master, Principal Investigator — Guizhou Provincial Cancer Hospital
Locations (1):
- Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China